CLINICAL TRIAL: NCT06026670
Title: Optimal Positive End-Expiratory Pressure in Robotic-Assisted Thoracic Surgery
Acronym: PEEP-RATS
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2023/0147
Record Dates: First submitted 2023-07-25; First posted 2023-09-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-07

CONDITIONS: Ventilator-Induced Lung Injury
Keywords: Optimal PEEP; Robotic-Assisted Thoracic Surgery.; Recruitment Maneuvers; Mechanical Ventilation; One-lung ventilation; Capnothorax; Positive End-Expiratory Pressure
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Minimally invasive thoracic surgery is increasingly popular. Recently, a new minimally invasive thoracic approach, robotic-assisted thoracic surgery (RATS) has been developed. RATS presents some advantages compared to VATS such as three-dimensional view of the surgical field, its precisions facilitates the navigation in difficult to access spaces and eliminates tremor which reduces learning curve and it may have a reduction of complications.

During RATS and differently from VATS, not only one lung ventilation (OLV) is needed but also a continuous tension capnothorax. CO2 insufflation with intrathoracic positive pressure has a potential negative impact on the cardiorespiratory physiology. Moreover, CO2 insufflation and one lung ventilation can produce ventilation induced lung injury which are related to pulmonary postoperative complications (PPC).

In order to reduce PPC and ventilation induced lung injury, lung protective strategies are used which reduce atelectrauma and overdistension. These strategies consist of three main pillars: use of low tidal volumes, performance of recruitment maneuvers and application of optimal positive end-expiratory pressure (PEEP).

However, optimal PEEP levels and actual effects of PEEP are not clear. Several clinical studies with one-lung ventilation have reported improved oxygenation and ventilation when an alveolar recruitment maneuver is performed with a standardized PEEP of 5 to 10 cm·H2O. Nevertheless, other studies observe during one-lung ventilation improvements in oxygenation and lung mechanics with individualized PEEP determined by using a PEEP decrement titration trial after an alveolar recruitment maneuver. The effect of a tension capnothorax during RATS may modify pulmonary compliance and optimal PEEP may be different from patients having VATS resection.

Even though both methods are habitual in the clinical practice, there are no studies of the effect of an alveolar recruitment maneuver with individualized PEEP during one-lung ventilation in Robotic-Assisted Thoracic Surgery (RATS). The investigators hypothesized that such a procedure would improve oxygenation and lung mechanics during one-lung ventilation in RATS compared with the establishment of a standardized PEEP. The investigators perform a descriptive observational prospective study to test this hypothesis.

DETAILED DESCRIPTION:
Minimally invasive thoracic surgery is increasingly popular thanks to its potential benefits, including less pain, reduced surgical stress and systemic inflammatory response and reduced length of stay. In fact, video-assisted thoracoscopic surgery (VATS), is recommended for lung resection in early stages in ERAS Guidelines. Recently, a new minimally invasive thoracic approach, robotic-assisted thoracic surgery (RATS) has been developed. Its main indications are lung resection, diaphragmatic repair, esophagectomy and resection of mediastinal tumor. RATS presents some advantages compared to VATS such as three-dimensional view of the surgical field, its precisions facilitates the navigation in difficult to access spaces, it improves work ergonomics and eliminates tremor which reduces learning curve and it may have a reduction of complications.

During RATS and differently from VATS, not only one lung ventilation (OLV) is needed but also a continuous tension capnothorax. Intrathoracic CO2 insufflation aims both to retract tissues and expand the surgical field which gives a better view of intrathoracic structures but also to facilitate anatomical dissection. Nevertheless, CO2 insufflation with intrathoracic positive pressure has a potential negative impact on the cardiorespiratory physiology: it may increase respiratory airway pressure, it may cause hypercapnia and respiratory acidosis and can compromise the hemodynamics induced by the compression of the mediastinal vessels. Moreover, CO2 insufflation and one lung ventilation can produce ventilation induced lung injury which are related to pulmonary postoperative complications (PPC).

In order to reduce PPC and ventilation induced lung injury, lung protective strategies are used which reduce atelectrauma and overdistension. These strategies consist of three main pillars: use of low tidal volumes, performance of recruitment maneuvers and application of optimal positive end-expiratory pressure (PEEP).

However, optimal PEEP levels and actual effects of PEEP are not clear. Several clinical studies with one-lung ventilation have reported improved oxygenation and ventilation when an alveolar recruitment maneuver is performed with a standardized PEEP of 5 to 10 cm·H2O. Nevertheless, other studies observe during one-lung ventilation improvements in oxygenation and lung mechanics with individualized PEEP determined by using a PEEP decrement titration trial after an alveolar recruitment maneuver. The effect of a tension capnothorax during RATS may modify pulmonary compliance and optimal PEEP may be different from patients having VATS resection.

Even though both methods are habitual in the clinical practice, there are no studies of the effect of an alveolar recruitment maneuver with individualized PEEP during one-lung ventilation in Robotic-Assisted Thoracic Surgery (RATS). The investigators hypothesized that such a procedure would improve oxygenation and lung mechanics during one-lung ventilation in RATS compared with the establishment of a standardized PEEP. The investigators perform a descriptive observational prospective study to test this hypothesis.

An individualized open lung approach which will consist in an alveolar recruitment maneuver followed by a positive end-expiratory pressure adjusted to best respiratory system compliance will be performed before and after capnothorax establishment.

The main expected benefits will be improvement of oxygenation, ventilation and lung mechanics.

Recruitment maneuvers are part of daily practice during mechanical ventilation. During OLV, they are done systematically, but little is known of optimal PEEP after it. When performed correctly, considering its contraindications and appropriate monitoring they are safe technique (9)

This is a single center (Hospital Clínic de Barcelona), prospective, intraoperative descriptive study. The hypothesis is to demonstrate the change in individualized optimal PEEP before and after capnothorax during OLV and the improvement of ventilation and lung mechanics. The primary objective is to assess the improvement of oxygenation, ventilation and lung mechanics in patients ventilated with individualized PEEP during capnothorax.The secondary objectives is to report the incidence of associated perioperative complications. With the purpose of standardizing the optimal respiratory management of patients that undergo robotic-assisted thoracic surgery (RATS).

Based on previous studies, it was estimated that a total of 30 patients will be needed to detect at least a 10% of static compliance during the establishment of capnothorax in one-lung ventilation, with a 5% significance level and 80% power.

Candidates for this study will be identified at the scheduled visit, prior to surgery, with one of the anaesthetists of the Cardiothoracic Anaesthesia section of our hospital. This visit is usually carried several days or weeks before surgery. Once a potential participant has been identified, the main investigator (R.N.) will offer the possibility to explain the study during the same scheduled visit and they will also provide written information regarding our study. Those who, subsequently, express their potential desire to participate in the study will also be offered an informed consent sheet for their signature. For those still willing to consider their participation but not ready to decide whether to accept or not their inclusion as part of the study, a second visit will be done once the patient is admitted to the hospital the day before the surgery.

The inclusion criteria are patients with ASA physical status I to III admitted to Hospital Clínic de Barcelona undergoing elective RATS lung resection who agree to participate in the study and sign the written consent form.

The exclusion criteria are patients with age <18 years, ASA physical status IV, pneumonectomy, New York Heart Association III to IV, and preoperative hemoglobin <10 mg/dL will be excluded from the study. Moreover, patients in which recruitment maneuvers are contraindicated will also be excluded from the study. Contraindications for recruitment maneuvers are: history of pneumothorax, contralateral pulmonary bulla, hemodynamic instability, lung emphysema, COPD, bronchopleural fistula, acute cor pulmonale or intracranial hypertension .

Data will be inspected and tested for distribution according to Kolmogorove Smirnov test. Normally distributed data were compared between study arms using the unpaired T-student test, whereas non-normally distributed data were compared using the Mann Whitney U test. All data were summarised as mean or median as appropriate. Fisher's exact test was used for comparing categorical data.

All patients included in the study will be assigned an identification code. In a separated database, the main investigator will have the relation between the identification code and the patient's clinical record number. All investigators of the study will have access to the coded number database that will be stored in a shared Drive document, and the main investigator will be responsible for it. Both database will be stored 5 years after study completion.

Individual data, such as participant baseline medical conditions, type of surgery, respiratory parameters, results from arterial gasometries samples and postoperative pulmonary complications until the 7th day from the admission will be recorded in order to assess the benefit of optimal PEEP before and after capnothorax stablishment.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I to III
* Admitted to Hospital Clínic de Barcelona
* Undergoing elective RATS lung resection
* Who agree to participate in the study and sign the written consent form.

Exclusion Criteria:

* Patients with age <18 years
* ASA physical status IV
* Pneumonectomy
* New York Heart Association III to IV
* Preoperative hemoglobin <10 mg/dL will be excluded from the study.
* Patients in which recruitment maneuvers are contraindicated (history of pneumothorax, contralateral pulmonary bulla, hemodynamic instability, lung emphysema, COPD, bronchopleural fistula, acute cor pulmonale or intracranial hypertension).

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ASA physical status I to III admitted to Hospital Clínic de Barcelona undergoing elective RATS lung resection who agree to participate in the study and sign the written consent form
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Optimal PEEP | 4 hours
  Assess the improvement of oxygenation, ventilation and lung mechanics in patients ventilated with individualized PEEP during capnothorax.

SECONDARY OUTCOMES:
Perioperative complications | 7 days
  Report the incidence of associated perioperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ricard Navarro, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No